CLINICAL TRIAL: NCT01830309
Title: Clinical Study to Evaluate Food-Effect on Pharmacokinetics and Pharmacodynamics of Single Oral Dose of CJ-12420 in Healthy Male Subjects
Brief Title: Food-Effect on PK and PD of Single Oral Dose of CJ-12420 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_APA_102
Record Dates: First submitted 2013-03-29; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Food-Effect; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Drug: CJ-12420 200mg Period1: CJ-12420 under fed condition Period2: CJ-12420 under fasting condition
  Interventions: Drug: CJ-12420 200mg
- Sequence 2 (Experimental): Drug: CJ-12420 200mg Period1: CJ-12420 under fasting condition Period2: CJ-12420 under fed condition
  Interventions: Drug: CJ-12420 200mg

INTERVENTIONS:
Drug: CJ-12420 200mg — Period1: CJ-12420 200mg fed condition Period2: CJ-12420 200mg fasting condition
  Period1: CJ-12420 200mg fasting condition Period2: CJ-12420 200mg fed condition
  Other Names: CJ-12420

SUMMARY:
* Primary: To evaluate food effect on the pharmacokinetics (PK) of a single oral dose of CJ-12420 in healthy male subjects.
* Secondary

  * To explore food effect on the pharmacodynamics (PD) of single oral dose of CJ-12420 in healthy male subjects(PD/PK group)
  * To evaluate the safety of single oral dose of CJ-12420 in healthy male subjects under fed or fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 45 years old(inclusive)
* Body mass index (BMI) in the range of 19 to 28 kg/m2 and weighing at least 50 kg (inclusive)
* Medically healthy with no clinically significant vital signs (sitting position blood pressure, pulse rate)

  1. 90 mmHg ≤ systolic blood pressure ≤ 140 mmHg
  2. 50 mmHg ≤ diastolic blood pressure ≤ 95 mmHg
  3. 45 beats per minute ≤ pulse rate ≤ 95 beats per minute
* Understand the requirements of the study and voluntarily consent to participate in the study

Exclusion Criteria:

Subjects will be excluded from the study if there is evidence of any of the following criteria: Last three criteria will be applied ONLY to PD/PK group.

* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary,immunologic, psychiatric, musculoskeletal or cardiovascular disease or any other condition, which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results
* History of allergy or sensitivity to any drug, including any prior serious adverse reaction to PPIs (e.g. omeprazole, rabeprazole, lansoprazole)
* History of symptomatic GERD, erosive esophagitis, duodenal ulcer, gastric ulcer, Barrett's esophagus or Zollinger-Ellison syndrome, previous positive H. pylori

The following criteria will be applied ONLY to PD/PK group

* H.pylori positive, as determined by the urea breath test
* Urine cotinine test positive
* Subject who were unable to be applicable for pH meter catheter

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Geometric mean ratio and 90% CI for log-transformed AUClast | Blood sampling during 24 or 48 hrs after administration
Geometric mean ratio and 90% CI for log-transformed Cmax | Blood sampling during 24 or 48 hrs after administration

SECONDARY OUTCOMES:
time pH > 4 | 24 hour before and after IP administration

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Han S, Choi HY, Kim YH, Nam JY, Kim B, Song GS, Lim HS, Bae KS. Effect of Food on the Pharmacokinetics and Pharmacodynamics of a Single Oral Dose of Tegoprazan. Clin Ther. 2021 Aug;43(8):1371-1380. doi: 10.1016/j.clinthera.2021.06.007. Epub 2021 Jul 8. PMID 34246485